CLINICAL TRIAL: NCT03774758
Title: Circulating Tumor DNA for Risk Stratification in Lung Cancer Screening
Brief Title: Biomarkers for Risk Stratification in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Northern California Institute of Research and Education (Other); Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-22915; 176517 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nodule Solitary Pulmonary; Non-small Cell Lung Cancer
Keywords: Lung cancer screening; Biomarkers of lung cancer; Circulating tumor DNA; Low dose computed tomography of lung; Pulmonary nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — The goal of this study is to evaluate the ability of cell-free circulating tumor DNA (ctDNA) using Guardant Health's LUNAR technology to detect early stage in lung cancer as compared to healthy volunteers and those patients at high risk for lung cancer, but without a lung cancer diagnosis. ctDNA arises when DNA fragments are released into the bloodstream after cell death and is distinguished from non-cancerous cell-free DNA (cfDNA) by the presence of somatic alterations, e.g. mutations, gene amplifications, and fusions. In advanced stage non-small cell lung cancer (NSCLC), evaluation of ctDNA in plasma can be used detect the presence of resistance mutations and ultimately guide treatment while obviating the need for tissue biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort 1A: Benign nodule on screening CT: High-risk patients eligible for lung cancer screening but with negative radiographic findings on CT screening (Lung RADS ≤2).
  1. ≥30 pack-year history of cigarette smoking
  2. ≥55 years of age
  3. Current smoker or quit within the past 15 years
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay
- Cohort 1B: Incidental benign nodule: Patients with lung nodules ≥ 6 mm on routine (non-lung cancer screening) CT evaluation deemed suspicious for malignancy by initial physician judgment but not malignant by ≥2 years of radiographic stability and consensus clinical opinion.
  1- Age ≥40 years.
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay
- Cohort IC: Presumed lung cancer: Patients with lung cancer (histologically proven or presumed by consensus opinion of tumor board); prior to definitive therapy.
  1- Age ≥40 years.
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay
- Cohort 2A: Suspicious nodule: High-risk patients with newly diagnosed suspicious nodule of Lung RADS ≥3 on CT screening.
  1. ≥30 pack-year history of cigarette smoking
  2. ≥55 years of age
  3. Current smoker or quit within the past 15 years
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay
- Cohort 2B: Suspicious incidental nodule: Patients with newly diagnosed incidentally-found lung nodules ≥ 6 mm on routine CT evaluation deemed suspicious for malignancy by physician judgment.
  1- Age ≥40 years.
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay
- Cohort 2C: Post-treatment lung cancer: Patients with previously treated lung cancer (histologically proven or by consensus opinion); status-post completion of definitive therapy (resection +/- chemotherapy or SBRT with curative intent) within the previous year with no current evidence of disease.
  1- Age ≥40 years.
  Interventions: Diagnostic Test: Guardant Health ct-DNA LUNAR assay

INTERVENTIONS:
Diagnostic Test: Guardant Health ct-DNA LUNAR assay — Guardant Health is focused on conquering cancer by using its breakthrough blood-based assays, vast data sets, and advanced analytics. In 2016, it announced Project LUNAR, an effort to apply Guardant Health's technology platform to early detection, recurrence monitoring, and assessing minimal residual disease.
  Other Names: Liquid biopsy Using NGS to Assay high-Risk patients

SUMMARY:
This is a prospective observational study that will follow patients who undergo lung cancer screening at the San Francisco VA Medical Center, University of California, San Francisco (UCSF) Medical Center, and the San Francisco General Hospital. The proposed study will comprise of two primary populations to determine the ctDNA assay performance in a variety of clinical settings.

DETAILED DESCRIPTION:
Study objectives and statistical approaches to achieve those objectives are determined at the level of the populations described below:

Population 1: Sensitivity and Specificity Thresholding.

In this phase, the technical feasibility of the intended use case will be assessed in the intended use population relative to known cancer status as established by standard clinical methods. ctDNA samples from enrolled patients will be assessed in each of the following cohorts:

Cohort 1A: High-risk patients negative for lung cancer by CT screening and clinical follow-up.

Cohort 1B: Patients with lung nodules ≥6 mm by CT but negative for lung cancer by extended (3 years) CT screening follow-up.

Cohort 1C: Patients with lung cancer (histologically proven or by consensus tumor board opinion of ≥90% probability of cancer) prior to definitive therapy.

Population 2: Clinical Intended Use Performance. In this phase, the clinical performance of the ctDNA assay will be evaluated in patients with high clinical suspicion for lung cancer. ctDNA will be compared to the clinical diagnosis made according to the standard of care (e.g. biopsy, CT surveillance, etc.). ctDNA samples from enrolled patients will be assessed in each of the following cohorts:

Cohort 2A: High-risk patients newly positive (Lung imaging Reporting And Data System (Lung-RADS) >=3) by CT screening.

Cohort 2B: Patients with >= 6 mm lung nodules suspicious for lung cancer by treating physician judgment.

Cohort 2C: Patients with a personal history of lung cancer after completion of curative intent treatment but without evidence of recurrence.

Specific Aim 1: To estimate the ctDNA assay sensitivity and specificity requirements in the specific clinical use populations using patients with known non-small cell lung cancer status.

Specific Aim 2: To prospectively estimate the ctDNA assay clinical performance in the clinical application of interest.

ENDPOINTS

Primary Endpoints

Specific Aim 1: Estimation of the ctDNA assay's clinical sensitivity and specificity in patients with lung cancer as proven by histology or tumor board consensus opinion* and in patients with lung nodule ≥6 mm but without cancer as proven by extended CT screening follow-up**.

*Patients may be treated with curative-intent Stereotactic Body Radiotherapy (SBRT) without tissue confirmation IF pretest probability for lung cancer by tumor board consensus opinion is ≥90% and the biopsy risk is high.

**Extended CT screening follow-up defined by documentation of ≥3 years of radiographic stability and consensus clinical opinion.

Specific Aim 2: Estimation of the ctDNA assay's clinical predictive value relative to standard of care diagnostic work-up in suspicious nodule adjudication in both the high-risk and general populations (the clinical applications of interest).

Secondary Endpoints

* Correlation of the ctDNA assay performance with Lung-RADS radiographic criteria
* Correlation of Lung-RADS with disease truth defined by clinical follow up as the definite gold standard

Exploratory Endpoints

* Correlation of plasma and tissue genotyping results
* Correlation of the ctDNA assay with orthogonal reference technologies (e.g. ddPCR)
* Correlation of the ctDNA assay performance with histologic sub-type and clinical course (e.g. aggressive vs. indolent disease)
* Correlation of the ctDNA assay performance with clinical lung cancer risk factors
* Correlation of the ctDNA assay results pre-and post-resection
* Correlation of follow-up the ctDNA assay results and kinetics vs. clinical recurrence post-resection or radiotherapy
* Estimation of theoretical biopsy avoidance rate in clinical use population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Ability to understand and provide written informed consent
* Willingness to comply with study protocols and provide blood samples.
* Willingness to complete 3-year clinical follow up

Exclusion Criteria:

* Active non-cutaneous malignancy within the past 5 years as per medical record or patient report.
* Exclusion criteria for possible follow-up visit blood draw:
* Anemia - measured by hematocrit level of less than 30%, measured after the first blood draw.
* Malnourishment - determined by BMI less than 19. If subject has BMI greater or equal to 19, but has a history of malnourishment, study staff will measure albumin level of subject's blood after initial blood draw. Albumin level must be greater than 2.5 mg per deciliter, or subject will be excluded.
* Severe Chronic Obstructive Pulmonary Disease (COPD) - defined by Gold Stage IV.
* Unstable heart conditions - defined by stable or unstable angina, recent myocardial infarction (within the last 2 years), active congestive heart failure, ischemic cardiomyopathy, or history of complications because of previous blood donation.
* Liver cirrhosis.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study that will follow patients who undergo lung cancer screening at the San Francisco VA Medical Center, UCSF Medical Center, and the San Francisco General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2017-12-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of ct-DNA LUNAR Assay | Extended CT screening follow-up defined by documentation of ≥3 years of radiographic stability and/or consensus clinical opinion by tumor board.
  Estimation of the ctDNA assay's clinical sensitivity and specificity in patients with lung cancer as proven by histology or tumor board consensus opinion* and in patients with lung nodule ≥6 mm but without cancer as proven by extended CT screening follow-up**.
  *Patients may be treated with curative-intent Stereotactic Body Radiotherapy (SBRT) without tissue confirmation IF pretest probability for lung cancer by tumor board consensus opinion is ≥90% and the biopsy risk is high.
Prospective negative predictive value of ct-DNA LUNAR assay | Extended CT screening follow-up defined by documentation of ≥3 years of radiographic stability and/or consensus clinical opinion by tumor board.
  Estimation of the ctDNA assay's clinical predictive value relative to standard of care diagnostic work-up in suspicious nodule adjudication in both the high-risk and general populations (the clinical applications of interest).

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Arjomandi, M.D., Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No